CLINICAL TRIAL: NCT00338091
Title: Long-Term Renoprotection of Optimal Antiproteinuric Doses of Benazepril and Losartan in Chronic Renal Insufficiency
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROAD
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2006-06-20 (Estimated); Status verified 2002-01

CONDITIONS: Renal Insufficiency,Chronic; Disease Progression; Proteinuria; Dose-Response Relationship,Drug; ACE Inhibitor; Angiotensin II Type 1 Receptor Blockers
Keywords: Renal Insufficiency,Chronic; Disease Progression; Proteinuria; Dose-Response Relationship,Drug; Benazepril; Losartan
MeSH Terms: conditions — Renal Insufficiency, Chronic; Disease Progression; Proteinuria | interventions — benazepril; Losartan

INTERVENTIONS:
Drug: Benazepril
Drug: Losartan

SUMMARY:
The primary goal of the trial was to evaluate whether the optimal antiproteinuric doses of benazepril (an ACE inhibitor) or losartan (an ARB), as compared with their conventional doses, can safely improve the long-term renal outcome in nondiabetic patients with proteinuria and chronic renal insufficiency. The second aim was to compare the long-term renal protection between benazepril and losartan at similar clinical setting.

ELIGIBILITY:
Inclusion Criteria:

1. Serum creatinine concentration of 1.5 to 5.0 mg per deciliter (133 to 442 µmol/L)
2. Creatinine clearance of 20 to 70 ml per minute per 1.73m2, with variations of less than 30 percent in the three months before screening evaluation
3. nondiabetic renal disease
4. Persistent heavier proteinuria (defined by urinary protein excretion of more than 1.0 g per day for three or more months without evidence of urinary tract infection or overt heart failure [a New York Heart Association class of Ⅲ or Ⅳ])

Exclusion Criteria:

1. Immediate need for dialysis
2. Treatment with corticosteroids, non steroidal anti-inflammatory drugs, or immunosuppressive drugs
3. Hyper-or hypokalemia (serum potassium concentration 5.6 mmol per liter or more，or 3.5 mmol per liter or less)
4. Renovascular disease
5. Myocardial infarction or cerebrovascular accident in the year preceding the trial
6. Connective-tissue disease; and obstructive uropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Study Completion 2006-05

PRIMARY OUTCOMES:
The primary efficacy measure was the time to the first event of the composite endpoint of a doubling of the serum creatinine concentration, ESRD or death.

SECONDARY OUTCOMES:
Secondary endpoints included changes in urinary protein excretion rate and the progression of renal disease assessed by creatinine clearance and glomerular filtration rate as calculated by Modification of Diet in Renal Disease equation-4.

CONTACTS AND LOCATIONS:
Overall Officials: Fan Fan Hou, M.D.,Ph.D., Principal Investigator — Division of Nephrology, Nanfang Hospital,Southern Medical University,China
Locations (1):
- Renal Division, Nanfang Hospital,Southern Medical University, Guangzhou, Guangdong, China